CLINICAL TRIAL: NCT00286975
Title: Growing Future Physician Leaders: A Randomized, Controlled Trial of an Educational Intervention in Postgraduate Trainees
Brief Title: Growing Future Physician Leaders: A Randomized Trial of an Educational Intervention in Postgraduate Trainees
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Royal College of Physicians and Surgeons of Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MDLead:Patel et al.
Record Dates: First submitted 2006-02-01; First posted 2006-02-06 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2005-11

CONDITIONS: Leadership Skills and Knowledge in Postgraduate Trainees
Keywords: Leadership skills; Management skills; Postgraduate medical education

INTERVENTIONS:
Behavioral: Leadership development program educational intervention

SUMMARY:
Study objective: The objective of this trial was to determine the effectiveness of a Leadership Development Program (LDP) aimed at 1) establishing basic management knowledge and 2) promoting reflection of leadership skills.

Study design: Randomized, controlled, single-blind trial. Study participants: Senior postgraduate medical and surgical trainees at an urban university health care centre.

Methods: Eligible participants were randomized to either the LDP(intervention group) or to regular postgraduate training (control group). For ethical reasons, all participants assigned to the control group were offered the LDP at the end of the trial. The 1º outcome measure used was a knowledge-based written exam. The sample size was estimated on finding a 20% difference in mean test scores between groups. Participants' reflective capacity and higher order leadership role skills were tested through a personal learning project (PLP, 2º outcome measure).

DETAILED DESCRIPTION:
Study objective: The objective of this trial was to determine the effectiveness of a Leadership Development Program (LDP) aimed at 1) establishing basic management knowledge and 2) promoting reflection of leadership skills.

Study design: Randomized, controlled, single-blind trial. Study participants: Senior postgraduate medical and surgical trainees at an urban university health care centre.

Methods: Eligible participants were randomized to either the LDP(intervention group) or to regular postgraduate training (control group). For ethical reasons, all participants assigned to the control group were offered the LDP at the end of the trial. The 1º outcome measure used was a knowledge-based written exam. The sample size was estimated on finding a 20% difference in mean test scores between groups. Participants' reflective capacity and higher order leadership role skills were tested through a personal learning project (PLP, 2º outcome measure).

ELIGIBILITY:
Inclusion Criteria: Postgraduate trainees in PGY 3 or higher -

Exclusion Criteria: Program director does not allow participation

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Hema Patel, MD, MSc, FRCP, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Silva JAM, Mininel VA, Fernandes Agreli H, Peduzzi M, Harrison R, Xyrichis A. Collective leadership to improve professional practice, healthcare outcomes and staff well-being. Cochrane Database Syst Rev. 2022 Oct 10;10(10):CD013850. doi: 10.1002/14651858.CD013850.pub2. PMID 36214207